CLINICAL TRIAL: NCT07025460
Title: Darbepoetin Alfa Once Monthly Dosing Schedule Maintains Hemoglobin Concentration Comparable to Every 2 Weeks Dosing Schedule in Advanced Chronic Kidney Disease Patients Not on Dialysis: A Multicenter, Phase 4 Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Hoon Young Choi, Clinical Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2019-0358
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: This study uses a single-group, open-label design in which all enrolled participants receive the investigational intervention-subcutaneous administration of darbepoetin alfa once monthly. After a 12-week screening phase with biweekly dosing to confirm hemoglobin stability and dosing consistency, eligible participants are transitioned to once-monthly dosing for a 12-week evaluation period. There is no comparator or randomization. All participants receive the same treatment protocol, and outcomes are assessed within this single cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Once-monthly darbepoetin alfa group (Experimental): Participants receive darbepoetin alfa administered subcutaneously once every 4 weeks for 12 weeks. Initial dose is based on prior month's cumulative dose. Dose adjustments are made based on hemoglobin levels to maintain Hb within 10.0-11.0 g/dL.
  Interventions: Drug: darbepoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — Participants receive darbepoetin alfa administered subcutaneously once every 4 weeks for 12 weeks during the evaluation phase. Dose adjustments are made to maintain hemoglobin levels within 10.0-11.0 g/dL.

SUMMARY:
This open-label, multicenter, single-arm phase 4 trial evaluated the efficacy and safety of once-monthly subcutaneous administration of darbepoetin alfa (DARB) compared with biweekly dosing in Korean patients with non-dialysis chronic kidney disease (ND-CKD) and anemia.

Anemia in CKD is a major contributor to cardiovascular morbidity and mortality. Although DARB every-2-week dosing has been established as effective, once-monthly dosing may maintain Hb levels while improving patient adherence and reducing healthcare burden. No clinical data were previously available for the Korean population, which is rapidly aging and has a high prevalence of CKD.

Study Design:

A total of 65 patients entered a 12-week screening period during which they received DARB every 2 weeks. Of these, 40 patients met eligibility criteria (stable Hb ≥9.5 g/dL, <25% dose variation) and were enrolled into the 12-week evaluation phase with once-monthly DARB dosing. Dose adjustments were made based on Hb trends to maintain Hb within 10.0-11.0 g/dL. All 40 patients completed the study and were included in efficacy and safety analyses.

Primary Endpoint:

Proportion of participants maintaining Hb ≥10.0 g/dL at Week 25, assessed for non-inferiority with a prespecified margin of 0.2 g/dL.

Secondary Endpoints:

Mean Hb concentration during the evaluation phase (Weeks 13, 17, 21, and 25)

Response frequency

Proportion of patients with Hb <10 g/dL or >11 g/dL

Change in iron parameters (serum ferritin, transferrin saturation)

Total DARB dose administered

Requirement for oral iron supplementation

Incidence of adverse events and blood pressure changes

Eligibility Criteria:

Inclusion:

Age ≥19 years

Diagnosis of CKD not requiring dialysis

eGFR ≤45 mL/min/1.73m² (MDRD formula)

Mean Hb ≤11.5 g/dL during screening, with Hb ≥9.5 g/dL

Stable DARB dosing during screening (<25% variation)

Ferritin ≥100 µg/L or transferrin saturation (TSAT) >20%

Exclusion:

Non-CKD causes of anemia

Acute myocardial infarction or hospitalization for heart failure within the past 12 weeks

Hematologic diseases, active infection, or recent major surgery

RBC transfusion within 8 weeks prior to screening, or DARB >180 mcg in the month prior to enrollment

Uncontrolled hypertension

Active malignancy

Sample Size:

A total of 77 patients were planned for enrollment, accounting for an expected dropout rate of 20%. In practice, 65 patients entered screening, 40 patients were enrolled into the evaluation phase, and all 40 completed the study.

Safety Considerations:

No unexpected safety issues were identified. Blood pressure remained stable throughout the study. Potential risks such as cardiovascular complications and tumor progression were considered; patients with significant risk factors were excluded. All data were anonymized and securely protected.

Significance:

This study provides real-world evidence that once-monthly DARB is non-inferior to biweekly dosing for maintaining Hb in Korean patients with ND-CKD. Extending the dosing interval to monthly administration may improve patient adherence, reduce injection burden, and inform treatment strategies for anemia management in Korea's aging CKD population.

DETAILED DESCRIPTION:
Study Design and Procedures

This was a prospective, open-label, multicenter, single-arm phase 4 clinical trial designed to evaluate the efficacy and safety of once-monthly subcutaneous darbepoetin alfa (DARB) compared with the established biweekly dosing schedule in Korean patients with anemia secondary to non-dialysis chronic kidney disease (ND-CKD).

Study Flow Summary

Screening Phase (Week -12 to 0):

A total of 65 patients received DARB every 2 weeks for 12 weeks. Eligibility required stable Hb levels (≥9.5 g/dL) with <25% dose variation during this period.

Enrollment (Week 0):

Forty patients who met all inclusion criteria and no exclusion criteria were enrolled into the evaluation phase and switched to once-monthly DARB dosing.

Evaluation Phase (Week 1 to 12):

Patients received once-monthly DARB for 12 weeks with predefined dose adjustments to maintain Hb within 10.0-11.0 g/dL.

Follow-up Visits:

Assessments were performed at Weeks 13, 17, 21, and 25.

Dosing Schedule

Initial monthly dose was based on the cumulative biweekly dose administered during the final month of the screening phase.

Dose titration rules:

Hb <10.0 g/dL → increase to next higher dose

Hb 10.0-11.0 g/dL → maintain current dose

Hb >11.0-12.0 g/dL → reduce to next lower dose

Hb >12.0 g/dL → temporarily withhold, reinitiate at lower dose once Hb ≤12.0 g/dL

Available doses: 20, 30, 40, 60, and 120 mcg (prefilled syringes).

Laboratory and Clinical Assessments

Hemoglobin, serum iron, ferritin, transferrin saturation (TSAT), TIBC, creatinine, eGFR (MDRD), and blood pressure were measured at scheduled visits.

Safety assessments included adverse event monitoring, physical examinations, and routine laboratory tests.

Statistical Considerations

Primary endpoint: Proportion of patients maintaining Hb ≥10.0 g/dL at Week 25, analyzed for non-inferiority with a prespecified margin of 0.2 g/dL.

Secondary endpoints: Mean Hb, iron parameters, response frequency, total DARB dose, oral iron requirements, and safety outcomes including adverse events and blood pressure changes.

Analysis sets:

Full Analysis Set (FAS): All 40 enrolled patients who received ≥1 dose and had ≥1 post-baseline Hb measurement.

Per-Protocol (PP) Set: Patients in the FAS without major protocol deviations who completed the study.

Missing data were imputed using Next Observation Carried Backward (NOCB).

Study Completion

Of the 65 patients screened, 40 entered the evaluation phase and all 40 completed the study, allowing full assessment of efficacy and safety outcomes.

Significance

This trial demonstrates that once-monthly darbepoetin alfa is non-inferior to biweekly dosing for maintaining hemoglobin in Korean patients with ND-CKD. These findings support the feasibility of extending the dosing interval to monthly administration, potentially improving adherence and reducing treatment burden in real-world practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Diagnosis of chronic kidney disease (CKD) not requiring dialysis
* Estimated glomerular filtration rate (eGFR) ≤ 45 mL/min/1.73 m² (calculated using the MDRD formula)
* Mean hemoglobin (Hb) concentration ≤ 11.5 g/dL during the screening period Hb concentration ≥ 9.5 g/dL during the screening period Stable DARB dosing during screening (defined as <25% variation in dose)
* Serum ferritin ≥ 100 µg/L or transferrin saturation (TSAT) > 20%
* Serum vitamin B12 and folate levels above the lower limit of normal (screening only) Provided written informed consent prior to any study-specific procedures

Exclusion Criteria:

* Planned kidney transplantation or prior kidney transplant
* Uncontrolled hypertension (systolic BP > 180 mmHg or diastolic BP > 110 mmHg) Acute myocardial infarction or hospitalization for heart failure within the past 12 weeks
* Serum parathyroid hormone (PTH) > 1500 pg/mL (screening only) Active systemic infection
* Diagnosed hematologic diseases (e.g., sickle cell anemia, myelodysplastic syndrome, leukemia, multiple myeloma, hemolytic anemia)
* Major surgery within 12 weeks prior to screening (excluding vascular access surgery)
* Red blood cell transfusion within 8 weeks before screening or during the study period
* Use of any investigational drug or medical device within 30 days prior to screening or during the study
* Active malignancy not in remission
* Total darbepoetin alfa dose > 180 mcg in the month prior to enrollment

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2026-01-18 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants maintaining hemoglobin (Hb) ≥10.0 g/dL at Week 25 | Week 25 (end of 12-week evaluation phase)
  The primary endpoint is the proportion of participants whose hemoglobin (Hb) concentration is maintained at or above 10.0 g/dL at Week 25 following once-monthly subcutaneous administration of darbepoetin alfa. Non-inferiority was assessed using a prespecified margin of 0.2 g/dL.

SECONDARY OUTCOMES:
Hemoglobin profile during the evaluation phase | Weeks 13, 17, 21, and 25
  Mean hemoglobin concentration at each visit and the proportion of participants outside the target range (Hb <10 g/dL or >11 g/dL).
Iron metabolism and treatment requirements | Weeks 13-25
  Changes in serum ferritin and transferrin saturation (TSAT), total darbepoetin alfa dose administered, and proportion of participants requiring oral iron supplementation.
Safety outcomes | Weeks 1-25
  Incidence, type, and severity of adverse events (AEs), and changes in systolic and diastolic blood pressure during the evaluation phase.

CONTACTS AND LOCATIONS:
Locations (1):
- Institutional Review Board, Gangnam Severance Hospitial Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hertel J, Locay H, Scarlata D, Jackson L, Prathikanti R, Audhya P. Darbepoetin alfa administered every other week maintains hemoglobin levels over 52 weeks in patients with chronic kidney disease converting from once-weekly recombinant human erythropoietin: results from simplify the treatment of anemia with Aranesp (STAAR). Am J Nephrol. 2006;26(2):149-56. doi: 10.1159/000092852. Epub 2006 Apr 21. PMID 16636531
- [Background] Roger SD, Kolmakova E, Fung M, Malecki R, Vinhas J, Dellanna F, Thomas M, Manamley N, Ferenczi S. Darbepoetin alfa once monthly corrects anaemia in patients with chronic kidney disease not on dialysis. Nephrology (Carlton). 2014 May;19(5):266-74. doi: 10.1111/nep.12214. PMID 24506498